CLINICAL TRIAL: NCT07145944
Title: To Explore the Application Value of Magnetic Resonance Imaging in Noninvasive Quantitative Evaluation of Graft Function and Systemic Metabolism After Renal Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhen Li, Professor, Tongji Hospital
Other Study IDs: TJ-IRB202411041
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Kidney Transplant Failure and Rejection; Transplantation, Kidney; Kidney Transplant Dysfunction
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- renal allograft patients: renal allograft patients

SUMMARY:
At present, renal biopsy is the gold standard for evaluating the pathology of renal transplants, but it is invasive and has the risk of serious complications; and the sampled tissue is only a small part of the kidney, which is prone to sampling bias and lacks reliable and comprehensive detection results. Therefore, it is an urgent problem to develop a non-invasive dynamic detection method for renal insufficiency and transplanted kidney.

With the continuous development and updating of technology, imaging provides a new way for non-invasive evaluation of renal allograft pathology including rejection reaction, acute renal allograft injury, viral infection, etc. MRI technology has developed the diagnosis of renal allograft rejection, fibrosis and other renal allograft dysfunction from macroscopic simple biomorphological changes to microscopic complex pathophysiological changes due to its high resolution of soft tissue and its ability to perform multi-parameter analysis.

In recent years, under the background of precision medicine, artificial intelligence technologies such as radiomics and machine learning are rapidly becoming very promising auxiliary tools in the evaluation of transplanted kidney images. They can extract and learn features in images with high throughput, make greater use of information that cannot be recognized by human eyes in medical images, and realize disease diagnosis, prognosis evaluation, and curative effect prediction by establishing models. However, most of the current research is in the preliminary stage. There are few evaluation studies on kidney transplantation. It is believed that with the continuous improvement of algorithms and optimization of models, radiomics and machine learning will make great progress, which will promote the development of individualized and precise medicine for patients with renal insufficiency to a certain extent.

DETAILED DESCRIPTION:
At present, renal biopsy is the gold standard for evaluating the pathology of renal transplants, but it is invasive and has the risk of serious complications; and the sampled tissue is only a small part of the kidney, which is prone to sampling bias and lacks reliable and comprehensive detection results. Therefore, it is an urgent problem to develop a non-invasive dynamic detection method for renal insufficiency and transplanted kidney.

With the continuous development and updating of technology, imaging provides a new way for non-invasive evaluation of renal allograft pathology including rejection reaction, acute renal allograft injury, viral infection, etc. MRI technology has developed the diagnosis of renal allograft rejection, fibrosis and other renal allograft dysfunction from macroscopic simple biomorphological changes to microscopic complex pathophysiological changes due to its high resolution of soft tissue and its ability to perform multi-parameter analysis.

In recent years, under the background of precision medicine, artificial intelligence technologies such as radiomics and machine learning are rapidly becoming very promising auxiliary tools in the evaluation of transplanted kidney images. They can extract and learn features in images with high throughput, make greater use of information that cannot be recognized by human eyes in medical images, and realize disease diagnosis, prognosis evaluation, and curative effect prediction by establishing models. However, most of the current research is in the preliminary stage. There are few evaluation studies on kidney transplantation. It is believed that with the continuous improvement of algorithms and optimization of models, radiomics and machine learning will make great progress, which will promote the development of individualized and precise medicine for patients with renal insufficiency to a certain extent.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients with MR examination after kidney transplantation;

  (2) Age/gender: unlimited;

  (3) Patients who voluntarily participate in clinical trials and sign written subject informed consent

Exclusion Criteria:

- (1) Patients with pacemakers, unknown materials, metal implants, neurostimulators, claustrophobia, etc.

(2) Patients who cannot tolerate adequate breath-holding for adequate MR examination;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: renal allograft patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2031-12-12 (Estimated)

PRIMARY OUTCOMES:
ESKD | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  The patient reaches CKD stage 5 and the glomerular filtration rate is less than 15 ml/min